CLINICAL TRIAL: NCT06879535
Title: ESTUDIO DE APLICACIÓN DE ESCALAS PARA VALORACIÓN SINTOMÁTICA DEL SÍNDROME DE COVID PERSISTENTE
Brief Title: Long-term Symptomatic Follow-up of Patients with Long COVID Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Andrés Carrascosa Gil, Médico Licenciado Especialista en Anestesiología y Reanimación, Hospital del Rio Hortega
Other Study IDs: 21-PI197
Record Dates: First submitted 2025-03-12; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
Keywords: Long COVID; Long-term follow-up; Symptoms; Scales
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Patients diagnosed with long COVID
- Controls: Patients who have had COVID acute infection without developing long COVID

SUMMARY:
The goal of this observational study is to learn about the long-term evolution of long COVID.

The main question it aims to answer is:

Does the main symptoms of the patients diagnosed with long COVID aproximate to those of patients who have had COVID acute infection without devoloping long COVID? Participants will answer mailed survey questions about their main symptons.

DETAILED DESCRIPTION:
Scales, indexes and questionnaires were mailed to 40 patients with long COVID to evaluate their main symptoms. Fatigue, emotional disorders, sleep disorders, cognitive impairments, dyspnea, physical activity, quality of life and pain were analyzed. The patients were reassessed after three years. The same scales, indexes and questionnaires were also sent to a control group of 40 volunteers of the same age and sex as the cases.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old and younger than 75 years old
* patients who accepted to participate in the study
* patients who have had COVID acute infection
* patients who have long COVID (cases)

Exclusion Criteria:

* patients who refused to participate in the study at any time of the study
* patients whose diagnosis of long COVID was revoked during the study (cases)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with long COVID who have been attended at the Internal Medicine Department at the Hospital Universitario Río Hortega from Valladolid
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Fatigue | From enrollment to three years later
  MFIS scale
Emotional disorders | From enrollment to three years later
  HADS scale
Sleep disorders | From enrollment to three years later
  PSQI
Cognitive impairments | From enrollment to three years later
  MFE-30
Dyspnea | From enrollment to three years later
  mMRC
Physical activity | From enrollment to three years later
  GPAQ
Quality of life (healthcare) | From enrollment to three years later
  SF-36
Pain (healthcare) | From enrollment to three years later
  EGDC

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Río Hortega, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided